CLINICAL TRIAL: NCT04342442
Title: Investigation of Novel Targetable Kinases in Steroid-refractory Acute Graft-versus-host Disease
Brief Title: Identification of Novel Targetable Kinases in SR-a GvHD
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Director of Division of Tumor Immunology, University of Freiburg
Other Study IDs: KIN-SR-GvHD
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Graft Versus Host Disease
Keywords: Steroid-refractory GvHD; Myeloid cells; Allogeneic hematopoietic cell transplantation (allo-HCT)
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Steroid-refractory a GvHD: Analysis of peripheral blood and intestinal biopsies of patients suffering from steroid-refractory a GvHD
- Steroid-responsive a GvHD: Analysis of peripheral blood and intestinal biopsies of patients suffering from steroid-responsive a GvHD

SUMMARY:
In this study, the investigators aim to identify novel targetable kinases in SR-a GvHD patient samples and investigate their role in different immune cell subtypes.

DETAILED DESCRIPTION:
Corticosteroids are the first-line treatment of a GvHD, however many patients do not respond to corticosteroids. Patients with steroid-refractory a GvHD (SR-a GVHD) have a low 1-year survival rate. In this study, the investigators aim to identify and validate novel targetable kinases in SR-a GvHD patient peripheral blood mononuclear cells (PBMCs) by using a kinase-specific proteomic approach, and thereafter to investigate the role of the identified kinases in different immune cell subtypes by analyzing biopsies taken from SR- a GvHD patients.

ELIGIBILITY:
Inclusion Criteria:

* allo-transplanted
* confirmed diagnosis of a GvHD
* age ≥ 18 years
* peripheral blood samples and biopsies available
* written informed consent
* ability to understand the nature of the study and the study-related procedures and to comply with them

Exclusion Criteria:

* age < 18 years
* lack of informed consent
* patients that cannot be classified in one of the 2 groups (steroid-refractory, steroid-responsive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute GvHD, steroid-refractory or steroid-responsive
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of differentially regulated kinases | 3 years
  Bead-based Kinase Assay enrichment (Knet beads) of PBMC lysates

SECONDARY OUTCOMES:
Analysis of protein expression | 3 years
  Analysis of PBMC lysates by western blot
Analysis of immune cell subtype | 3 years
  Immunohistochemistry of intestinal biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zeiser, Prof. Dr., Principal Investigator — University Medical Center Freiburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeiser R, Burchert A, Lengerke C, Verbeek M, Maas-Bauer K, Metzelder SK, Spoerl S, Ditschkowski M, Ecsedi M, Sockel K, Ayuk F, Ajib S, de Fontbrune FS, Na IK, Penter L, Holtick U, Wolf D, Schuler E, Meyer E, Apostolova P, Bertz H, Marks R, Lubbert M, Wasch R, Scheid C, Stolzel F, Ordemann R, Bug G, Kobbe G, Negrin R, Brune M, Spyridonidis A, Schmitt-Graff A, van der Velden W, Huls G, Mielke S, Grigoleit GU, Kuball J, Flynn R, Ihorst G, Du J, Blazar BR, Arnold R, Kroger N, Passweg J, Halter J, Socie G, Beelen D, Peschel C, Neubauer A, Finke J, Duyster J, von Bubnoff N. Ruxolitinib in corticosteroid-refractory graft-versus-host disease after allogeneic stem cell transplantation: a multicenter survey. Leukemia. 2015 Oct;29(10):2062-8. doi: 10.1038/leu.2015.212. Epub 2015 Jul 31. PMID 26228813
- [Background] Hulsdunker J, Ottmuller KJ, Neeff HP, Koyama M, Gao Z, Thomas OS, Follo M, Al-Ahmad A, Prinz G, Duquesne S, Dierbach H, Kirschnek S, Lammermann T, Blaser MJ, Fife BT, Blazar BR, Beilhack A, Hill GR, Hacker G, Zeiser R. Neutrophils provide cellular communication between ileum and mesenteric lymph nodes at graft-versus-host disease onset. Blood. 2018 Apr 19;131(16):1858-1869. doi: 10.1182/blood-2017-10-812891. Epub 2018 Feb 20. PMID 29463561
- [Background] Zeiser R, Blazar BR. Acute Graft-versus-Host Disease - Biologic Process, Prevention, and Therapy. N Engl J Med. 2017 Nov 30;377(22):2167-2179. doi: 10.1056/NEJMra1609337. No abstract available. PMID 29171820
- [Background] Schwab L, Goroncy L, Palaniyandi S, Gautam S, Triantafyllopoulou A, Mocsai A, Reichardt W, Karlsson FJ, Radhakrishnan SV, Hanke K, Schmitt-Graeff A, Freudenberg M, von Loewenich FD, Wolf P, Leonhardt F, Baxan N, Pfeifer D, Schmah O, Schonle A, Martin SF, Mertelsmann R, Duyster J, Finke J, Prinz M, Henneke P, Hacker H, Hildebrandt GC, Hacker G, Zeiser R. Neutrophil granulocytes recruited upon translocation of intestinal bacteria enhance graft-versus-host disease via tissue damage. Nat Med. 2014 Jun;20(6):648-54. doi: 10.1038/nm.3517. Epub 2014 May 18. PMID 24836575